CLINICAL TRIAL: NCT02350582
Title: e-CUIDACHEMO: Telerehabilitation During Chemotherapy in Breast Cancer Patients
Brief Title: e-CUIDACHEMO: Telerehabilitation During Chemotherapy in Breast Cancer
Acronym: e-CUIDACHEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Health Service of Andalucia (Other Government)
Responsible Party: Principal Investigator, Manuel Arroyo Morales, Associate Profesor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SAS-0457-2010
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; telerehabilitation; strength; fatigue; quality of life
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telerehabilitation (Experimental): Resistence and endurance exercise adapted to individual requeriment using internet to monitor progression during chemotherapy treatment. Telerehabilitation eCUIDATE system
  Interventions: Device: Telerehabilitation eCUIDATE system
- Control group (No Intervention): usual care offered to patients during chemotherapy treatment

INTERVENTIONS:
Device: Telerehabilitation eCUIDATE system — Resistence and endurance exercise adapted to individual requeriment during chemotherapy
  Arms: Telerehabilitation

SUMMARY:
Patients with breast cancer undergo a series of psiclofisicas alterations during cancer treatment, chemotherapy phase being one of the more aggressive ete effect. These changes reduce the quality of life and result in a loss of physical health-related condition. Studies have shown that the practice of physical exercise and rehabilitation strategies enhance or attenuate the impact of chemotherapy on quality of life of patients. At present, technological development from telerehabilitación systems is a promising strategy that enables fast and efficient communication between health professionals and patients, especially at this stage of the disease where the patient may encounter difficulties in matching measures improving their lifestyle with aggressive medical treatment.

To carry out this study a controlled study masked, parallel-group done were conducted usual care control group and an intervention based on a web system telerehabilitación to improve the physical condition associated with health and performed quality of life.

DETAILED DESCRIPTION:
The CUIDATE group will identify impairments of participants at baseline assessment. The aims based on weekly improvements will be set to facilitate the final goal. After each training session there will be feedback between the participant and the CUIDATE group to change or improve any exercise or activity. This feedback will allow to us to select adequate exercises and levels of difficulty. As a result, a modifiable personal training will be assigned to each one focusing on cardio-respiratory, mobility, and endurance performance through online system rehabilitation (using written instructions, HD videos, and audio files).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, II, or IIIA breast cancer
* Medical clearance of participation
* Access to the Internet
* Basic ability to use a computer or living with someone who has this ability
* In chemotherapy treatment at present moment;
* Have interest in improving lifestyle: fitness level
* Have signed informed consent

Exclusion Criteria:

* Chronic disease or orthopedic issues that would interfere with ability to participate in a physical activity program;

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2015-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory capacity | 1 day
  Distance in meters in 6 minutes walking test

SECONDARY OUTCOMES:
Abdominal endurance strength | 1 day
  Abdominal resistance using curl-up test
Lumbar extensor endurance strength | 1 day
  Lumbar extensor strength using dynamometer
Handgrip endurance strength | 1 day
  Handgrip endurance using isometric dynamometer
Cancer related fatigue | 2 days
  Piper Fatigue Scale
Cancer related pain | 2 days
  Brief Pain Inventory
Cancer related quality of life | 2 days
  EORTC Quality of life questionaire Core and Br23

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Arroyo-Morales, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of Health Sciences. University of Granada, Granada, Spain

REFERENCES:
- [Derived] Ariza-Garcia A, Lozano-Lozano M, Galiano-Castillo N, Postigo-Martin P, Arroyo-Morales M, Cantarero-Villanueva I. A Web-Based Exercise System (e-CuidateChemo) to Counter the Side Effects of Chemotherapy in Patients With Breast Cancer: Randomized Controlled Trial. J Med Internet Res. 2019 Jul 24;21(7):e14418. doi: 10.2196/14418. PMID 31342907